CLINICAL TRIAL: NCT01304160
Title: Phase I/II Study to Investigate the Role of Cyberknife Stereotactic Radiation Therapy (SBRT) Followed by Gemcitabine for Patients With Locally Advanced Pancreatic Cancer
Brief Title: Role of Cyberknife Stereotactic Radiation Therapy (SBRT) Followed by Gemcitabine for Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 09.153
Record Dates: First submitted 2011-02-21; First posted 2011-02-25 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2012-08

CONDITIONS: Pancreatic Cancer; Unresectable Pancreatic Cancer
Keywords: pancreatic cancer; stereotactic body radiotherapy; radiation; gemcitabine; locally advanced
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- strereotactic radiotherapy, gemcitabine (Experimental): stereotactic radiotherapy (30Gray in 5 fractions) followed by gemcitabine
  Interventions: Radiation: stereotactic body radiotherapy

INTERVENTIONS:
Radiation: stereotactic body radiotherapy — 30Gray in 5 fractions

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of stereotactic radiation therapy given in five fractions (30 Gray in 5 fractions) followed by gemcitabine in patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
The purpose of this phase I/II study is to evaluate the efficacy and toxicity of a different stereotactic body radiation therapy regimen combined with gemcitabine. In the present study, 5 daily fractions of 6 Gray will be given over two weeks. Stereotactic body radiation therapy will be given with the Cyberknife system. This treatment technique allows to give a higher dose to the tumor as compared to conventional external beam radiation while lowering the dose to the normal tissues around. This treatment system is also capable of following the motion that the pancreas assumes during respiration as well as during treatment. This enables us to reduce the margin of security and further reduce dose to surrounding normal tissue.

The primary objective of this study is to evaluate acute and chronic toxicity of this regimen of stereotactic radiation therapy followed by gemcitabine. Quality of life, local control and overall survival will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic Adenocarcinoma, histologically and/or cytologically proven
* Locally advanced pancreatic cancer, surgically non resectable
* No distant metastasis
* Work-up including medical history, physical exam, biochemistry, chest X-ray, CT-scan of abdomen and pelvis
* ECOG performance status : ≤ 2
* Primary tumor visible on CT-scan
* Maximum tumor diameter of 6 cm (including primary tumor and regional lymph nodes)
* White blood cell count > 3000 /uL, Neutrophils > 1500 /uL, Platelets > 100 000/uL, Hemoglobin > 95 mg/L, Total bilirubin < 1,5 normal limit, AST/ALT < 2,5 normal limit, normal creatinin
* ≥ 18 years of age
* Signed informed consent

Exclusion Criteria:

* Prior abdominal radiation therapy
* Connective tissue disease (scleroderma, lupus)
* Prior treatment for pancreatic cancer such as radiation therapy, chemotherapy or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | one year
  Acute and chronic toxicities will be evaluated according to the National Cancer Institute Common Toxicity Criteria version 3.0

SECONDARY OUTCOMES:
Quality of life | 3 monthly
  Quality of life will be evaluated with the EORTC QLQ-C30 questionnaire
Local control | 3 monthly
  Local control will be assessed with 3 monthly CT-scans of the abdomen. RECIST criteria will be used to evaluate local control.
overall survival | one and two year

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre Campeau, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada